IRB Protocol Number: 2020C0128 IRB Approval date: 5/30/2023

Version: 4

## The Ohio State University Combined Consent to Participate in **Research and HIPAA Research Authorization**

2 3

1

Re-Defining Frailty and Improving Outcomes Through

**Study Title: Prehabilitation (RIOT Trial)** 

**Principal Investigator:** Aslam Ejaz, MD

**Sponsor:** The Ohio State University

4 5

6

7

8

9

10

11

12

13

14

15

16

17

18

19

20

21

This is a consent form for research participation. It contains important information about this study and what to expect if you decide to participate. Please consider the information carefully. Feel free to discuss the study with your friends and family and to ask questions before making your decision whether or not to participate.

Your participation is voluntary. You may refuse to participate in this study. If you decide to take part in the study, you may leave the study at any time. No matter what decision you make, there will be no penalty to you and you will not lose any of your usual benefits. Your decision will not affect your future relationship with The Ohio State University. If you are a student or employee at Ohio State, your decision will not affect your grades or employment status.

- You may or may not benefit as a result of participating in this study. Also, as explained below, your participation may result in unintended or harmful effects for you that may be minor or may be serious depending on the nature of the research.
- You will be provided with any new information that develops during the study that may affect your decision whether or not to continue to participate. If you decide to participate, you will be asked to sign this form and will receive a copy of the form. You are being asked to consider participating in this study for the reasons explained below.

22 23 24

25

#### **Key Information About This Study**

The following is a short summary to help you decide whether or not to be a part of this study. More detailed information is listed later in this form.

26 27 28

29

This study is looking at a cancer patient's health before surgery, and if simple guided physical exercise before surgery will help to lower your risks and better your healing leading up to and following surgery.

- If you participate / if chosen for the exercise group, before surgery you may have your blood 32 33 drawn, be given simple exercises to do, and have possible follow up phone visits. There will be surveys to complete at appointments or through email after surgery for all that join. There 34
- 35 may also be a blood draw the day of surgery, and at your 1<sup>st</sup> first visit after surgery. We may

IRB Protocol Number: 2020C0128
IRB Approval date: 5/30/2023

Version: 4

also save some tissue samples from the pieces removed by your surgeon. Alternatively, if you participate, but are not chosen for the exercise group, you will still receive standard of care instructions, complete surveys and may have your blood drawn at the same time points, and again have tissues saved. The study lasts about 1 year.

#### 1. Why is this study being done?

 In an aging population, a pre-surgical (before surgery) risk check is done to decide if your cancer can be removed. Surgery provides the best hope for long-term survival among patients with abdominal/belly cancers (ex: localized pancreatic, liver, or gastric cancer -where the cancer is only in that organ). However, many of the patients who may have their pancreas, liver, or stomach removed will have problems after surgery. Though chemotherapy after surgery improves cancer-specific survival, many of patients who undergo abdominal cancer surgery will not receive any treatment due to the failure to heal from the surgery or surgery-related problems.

The usual way to check surgical risk is age and current diseases. This is not always accurate. Recently, the idea of frailty has been introduced as a better way to check for risk. Frailty is usually described as weakness related to aging, as well as illness and the ability to handle normal every day stress. Prehabilitation programs, or exercise programs before surgery, try to improve the medical and physical state of patients before surgery. This has not been well studied in people going through cancer surgery.

#### 2. How many people will take part in this study?

144 total (2 groups with 72 in each group)

## 3. What will happen if I take part in this study?

If you take part in the study, you will be given a study number, simple physical tests (like walking speed/6 minute walk, grip strength, timed up and go "TUG"), a few questions about your daily activities (Katz Index of Independence), feelings (CES-D), memory (mini-Cog), a quality of life questionnaire, as well as a short frailty survey to complete – these are a part of research.

A computer program will randomly, like flipping a coin, select if you will be in the no prehabilitation group or prehabilitation group. Prehabilitation, or prehab, is to help get stronger before an event, like surgery. (See Schedule of Activities on pg 4) The other group will be in the study as a non-prehab group, which means, not doing specific exercises before surgery, but continuing their daily activities as usual.

For those subjects in the non-prehab group, with no assigned exercises, you will receive presurgical information from your provider. For those randomized into the prehabilitation group, you will talk with a physical therapist. This is an expert in helping people that have limited

IRB Protocol Number: 2020C0128
IRB Approval date: 5/30/2023
Version: 4

activity or movement in their lives. They will give you low or moderate-high intensity home exercises to work on. These will be done at home during the time before your surgery, but you will have contact with a study team member for any questions. Some people may have trouble completing all the exercises at first, but we are hopeful that the more you try, the more you will be able to finish.

If assigned to the prehab group, the time at home (20-50 mins for 2-3 days/week) before your date for surgery, you will be doing the simple exercises given to you at the physical therapy session, and marking them on the exercise diary provided by physical therapy, in addition to any instructions provided by your care team. This one-time physical therapy session may take about 45-60 mins. A research team member will call you each week to check in on your progress and answer any questions you may have about the study. Those in the other group will follow any instructions as given by their care team only.

All enrolled subjects will have their blood drawn. Approximately 30cc or 1 tablespoon of blood may be drawn during your visit 0 (see below). This blood will be processed and stored until the end of the study, here at Ohio State, with your study number on it.

The day of surgery, blood may be drawn when other routine labs are drawn for all enrolled subjects as a part of the study. Also, a very small amount of your tissues, if not needed by pathology, will be taken. This is from the tissues already removed as a part of your surgery.

After surgery, all subjects will be scheduled to follow-up as part of your routine clinic care with your doctor. At this time as a part of this study, you will be asked to complete a quality of life questionnaire, and may have your blood drawn. If you were assigned the prehab group, you will-can return the exercise diary on the day of surgery, at one of your post-operative appointments or with the stamped, addressed envelope provided to you.

A study team member will review and collect medical information from all enrolled subjects, for basic information such as height, weight, type of surgery, complications, for example, but subjects will be identified by a study ID number.

124

125 126

127 128

129 130

#### Schedule of Activities

| | Visit 0 | Pre-operative / at home <sup>1</sup> | Phone visit <sup>1</sup> (s) | Visit 1<br>(Day of surgery) | Visit 2 -Week<br>2 Post-op | Visit 3-<br>Month 3<br>Post-op | Visit 4-<br>Month 6<br>Post-op | Visit 5-<br>Month 12<br>Post-op | End of Study |
|---|---|---|---|---|---|---|---|---|---|
| Informed Consent | X | | | | | | | | |
| Inclusion/exclusion criteria | X | | | | | | | | |
| History and Physical | X | | | | | | | | |
| FRAIL Questionnaire - Randomization | X | | | | | | | | |
| Subject interview / assessments | X | | | | | | | | |
| Physical Therapy consult | $X^1$ | | | | | | | | |
| Blood collection | X | | | X | X | | | | |
| Tissue collection – only what is already being removed from your usual surgery | | | | X | | | | | |
| Exercises | | X <sup>1</sup> | | | | | | | |
| Prehab check-in | | | $X^1$ | | | | | | |
| PROMIS survey | X | | | | X | X | X | X | X |
| 90-day morbidity assessed via Comprehensive<br>Complicaton Index (CCI) | | | | | | X | | | |
| AE Assessment | | | $X^1$ | | X | X | X | X | X |

1 -only if assigned to exercise

131 132 133 134 135 **Prehab check-in** at Phone visit – Follow-up on exercises, questions, AEs

 $AE-adverse\ event$ 

Post-op, post-operative/after surgery

Note: 90-day Morbidity = 3 month review of health status with a trusted guide 136

137 138

If you do not end up having surgery, you will be withdrawn from the study, and will be asked to complete the quality of life suvery (PROMIS).

139 140 141

#### 4. How long will I be in the study?

142143

144

145

Approximately 12 months for the entire study, however the exercise program (if you are in that group) will only be during the time between the first session with physical therapy and the day of your surgery. This could be about 2-4 weeks, but may vary depending on the date of your surgery.

146147148

#### 5. Can I stop being in the study?

149150

151

152

You may leave the study at any time. If you decide to stop participating in the study, there will be no penalty to you, and you will not lose any benefits to which you are otherwise entitled. Your decision will not affect your future relationship with The Ohio State University.

153154155

#### 6. What risks, side effects or discomforts can I expect from being in the study?

156157

158

With any exercise therapy program, there are slights risks including pulling or straining muscles, muscle soreness, shortness of breath, muscle tightness in your legs, arms, or abdomen, and in very rare cases dizziness or lightheadedness.

159 160 161

162

163

The doctor or study staff will take blood from a blood vessel in your arm by inserting a small needle. Possible side effects of taking blood this way may include tenderness, pain, and bruising at the site where the needle entered the arm, but this will be gone in a few days. Infection, lightheadedness, or fainting is rare.

164 165 166

There is a potential risk to your privacy. Every effort will be made to maintain your privacy, however this cannot be guaranteed.

167168169

#### 7. What benefits can I expect from being in the study?

170 171

You may or may not benefit from participating in this study. It is possible that exercise therapy, and the education may result in fewer complications following surgery. It is expected that this research will help others in the future.

173174175

172

## 8. What other choices do I have if I do not take part in the study?

176177

You may choose not to participate without penalty or loss of benefits to which you are otherwise entitled.

178179180

## 9. What are the costs of taking part in this study?

181 182

There is no cost for being in the study.

183

## 10. Will I be paid for taking part in this study?

You will not be paid for being in the study.

186 187 188

#### 11. What happens if I am injured because I took part in this study?

189 190

191

If you suffer an injury from participating in this study, you should notify the researcher or study doctor immediately, who will determine if you should obtain medical treatment at The Ohio State University Wexner Medical Center.

192 193 194

The cost for this treatment will be billed to you or your medical or hospital insurance. The Ohio State University has no funds set aside for the payment of health care expenses for this study.

196 197 198

195

#### 12. What are my rights if I take part in this study?

199 200

201

If you choose to participate in the study, you may discontinue participation at any time without penalty or loss of benefits. By signing this form, you do not give up any personal legal rights you may have as a participant in this study.

202 203 204

205

You will be provided with any new information that develops during the course of the research that may affect your decision whether or not to continue participation in the study.

206 207 208

You may refuse to participate in this study without penalty or loss of benefits to which you are otherwise entitled.

209 210 211

212

213

An Institutional Review Board responsible for human subjects research at The Ohio State University reviewed this research project and found it to be acceptable, according to applicable state and federal regulations and University policies designed to protect the rights and welfare of research participants.

214 215 216

#### 13. Will my de-identified information and bio-specimens be used or shared for future research?

217 218 219

Yes, they may be used or shared with other researchers without your additional informed consent.

220 221 222

## 14. Will my study-related information be kept confidential?

223 224

225

226

Efforts will be made to keep your study-related information confidential. However, there may be circumstances where this information must be released. For example, personal information regarding your participation in this study may be disclosed if required by state law.

227 228 229

Also, your records may be reviewed by the following groups:

IRB Protocol Number: 2020C0128
IRB Approval date: 5/30/2023
Version: 4

• Office for Human Research Protections or other federal, state, or international regulatory agencies;

- U.S. Food and Drug Administration;
- The Ohio State University Institutional Review Board or Office of Responsible Research Practices;
- The sponsor supporting the study, their agents or study monitors; and
- Your insurance company (if charges are billed to insurance).

236237238

230

231

232

233

234

235

If we find information that significantly impacts your health, we will share it with you, at your next appointment with your physician.

239240241

242

243

244

245

We will work to make sure that no one sees your survey responses without approval. But, because we are using the Internet, there is a chance that someone could access your online responses without permission. In some cases, this information could be used to identify you. Your data will be protected with a code to reduce the risk that other people can view the responses.

246247248

# 15. HIPAA AUTHORIZATION TO USE AND DISCLOSE INFORMATION FOR RESEARCH PURPOSES

249250

#### I. What information may be used and given to others?

251252

255

256

257

258

259

260

261

- Past and present medical records;
- Past and present nResearch records;
  - Records about phone calls made as part of this research;
  - Records about your study visits;
    - Information that includes personal identifiers, such as your name, or a number associated with you as an individual;
    - Information gathered for this research about:

Physical exams

Laboratory, x-ray, and other test results

Diaries and questionnaires

262263264

#### II. Who may use and give out information about you?

265266

Researchers and study staff.

267268

#### III. Who might get this information?

269270

271

- The sponsor of this research. "Sponsor" means any persons or companies that are:
  - working for or with the sponsor; or
  - owned by the sponsor.

• Authorized Ohio State University staff not involved in the study may be aware that you are participating in a research study and have access to your information;

• If this study is related to your medical care, your study-related information may be placed in your permanent hospital, clinic, or physician's office record;

IV Vousins

#### IV. Your information may be given to:

278279280

281

282

283

284

285

286

273

274

275

276277

• The U.S. Food and Drug Administration (FDA), Department of Health and Human Services (DHHS) agencies, and other federal and state entities;

• Governmental agencies in other countries;

- Governmental agencies to whom certain diseases (reportable diseases) must be reported; and
- The Ohio State University units involved in managing and approving the research study including the Office of Research and the Office of Responsible Research Practices.

287288

#### V. Why will this information be used and/or given to others?

289290

• To do the research;

291292

• To study the results; and

293294

• To make sure that the research was done right.

295296

## VI. When will my permission end?

297 298 There is no date at which your permission ends. Your information will be used indefinitely. This is because the information used and created during the study may be analyzed for many years, and it is not possible to know when this will be complete.

299300301

## VII. May I withdraw or revoke (cancel) my permission?

302 303

304

305

306

307

308

Yes. Your authorization will be good for the time period indicated above unless you change your mind and revoke it in writing. You may withdraw or take away your permission to use and disclose your health information at any time. You do this by sending written notice to the researchers. If you withdraw your permission, you will not be able to stay in this study. When you withdraw your permission, no new health information identifying you will be gathered after that date. Information that has already been gathered may still be used and given to others.

309310311

# VIII. What if I decide not to give permission to use and give out my health information?

IRB Protocol Number: 2020C0128
IRB Approval date: 5/30/2023

Version: 4

Then you will not be able to be in this research study and receive research-related 314 treatment. However, if you are being treated as a patient here, you will still be able to 315 316 receive care. 317 IX. Is my health information protected after it has been given to others? 318 319 There is a risk that your information will be given to others without your permission. Any 320 information that is shared may no longer be protected by federal privacy rules. 321 322 X. May I review or copy my information? 323 324 Signing this authorization also means that you may not be able to see or copy your study-325 related information until the study is completed. 326 327 328 16. Who can answer my questions about the study? 329 330 331 For questions, concerns, or complaints about the study, or if you feel you have been harmed as a result of study participation, you may contact Aslam Ejaz, MD, MPH at (614) 332 614-293-7171. 333 334 For questions related to your privacy rights under HIPAA or related to this research 335 authorization, please The Ohio State University Medical Center Privacy office at (614) 336 293-4477. 337 338 For questions about your rights as a participant in this study or to discuss other study-339 related concerns or complaints with someone who is not part of the research team, you 340 may contact the Office of Responsible Research Practices at 1-800-678-6251. 341 342 If you are injured as a result of participating in this study or for questions about a study-343

related injury, you may contact Aslam Ejaz, MD, MPH at (614) 614-293-7171.

345346

IRB Protocol Number: 2020C0128 IRB Approval date: 5/30/2023 Version: 4

| Signing the consent form | | |
|---|---|---|
| I have read (or someone has read to me) this participate in a research study. I have had the answered to my satisfaction. I voluntarily ag | e opportunity to ask questions and have have | |
| I am not giving up any legal rights by signing combined consent and HIPAA research authorized to the combined combined consent and HIPAA research authorized to the combined combined consent and HIPAA research authorized to the combined consent authorized to the combined cons | | |
| Printed name of participant | Signature of participant | |
| | Date and time | A |
| Printed name of person authorized to consent for participant (when applicable) | Signature of person authorized to consent for pa<br>(when applicable) | ırticipa |
| Relationship to the participant | Date and time | A |
| signature(s) above. There are no blanks in the to the participant or his/her representative. | is document. A copy of this form has bee | en giv |
| Printed name of person obtaining consent | Signature of person obtaining consent | |
| | Date and time | |
| Witness(es) - May be left blank if not req | | A |
| | quired by the IRB | A |
| Printed name of witness | Signature of witness | A |
| Printed name of witness | | |
| Printed name of witness Printed name of witness | Signature of witness | A |
| | Signature of witness Date and time | |